CLINICAL TRIAL: NCT05037916
Title: Comparison of Laser Speckle Contrast Imaging and Laser Doppler Imaging in Burn Patients
Acronym: COLA-B
Status: Completed | Type: Observational
Sponsor: Maasstad Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: L2019017 /NL66174.100.18
Record Dates: First submitted 2020-10-13; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2020-10

CONDITIONS: Laser Burn

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: laser speckle contrast imaging device — laser speckle contrast imaging device will be used for measurement of burn wound depth en to be compared to the golden standard the laser doppler imaging device

SUMMARY:
Timely and accurate estimation of the surface area and depth of a burn injury is essential for determining an appropriate treatment modality. Inappropriate or inadequate treatment may result in complications and increased societal costs. Burn depth is determined by subjective assessing the characteristics of burn injury. Some objective methods are available (e.g., biopsy and histology, thermography and laser doppler imaging), but these are cumbersome. In assessing burn wounds, laser Doppler imaging (LDI) which has a good correlation with histology, is currently the most widely used and validated noninvasive measurement tool. In addition, it is the only technique that has been approved by the U.S. Food and Drug Administration. However, the use of LDI is accompanied by some disadvantages. The current commercial available LDI device is rather costly, cumbersome and has a poor spatial resolution. Another laser-based technique, laser speckle contrast imaging (LSCI), works with a similar principle and might become an alternative for LDI. LSCI has some advantages over LDI such as higher spatial resolution, much easier to position, no valuable time wasted on setting up the instrument, easy to take several images of burns that have a large surface area and/or much curvature, faster measurements, fraction of the time needed for getting a high-quality measurement, able to follow changes in the perfusion in real time. In contrast to the LDI, the LSCI has not been validated in terms of a diagnostic tool for stratifying the severity of a burn (based on LDI color coding). Consequently, we will compare the LSCI with LDI to improve burn care by providing cheaper, faster and higher resolution imaging technique.

DETAILED DESCRIPTION:
After receiving adequate information and when informed consent is signed, patients are included. All patients receive usual care. Within 2-5 days post burn the LSCI and LDI are performed. Ideally, LDI is performed after 2 days, scanning up to 5 days is permitted when patients present later post burn or due to logistic reasons. The wounds are scanned by a trained research physician or nurse, during regular wound care.

8.4 Population base: Measurements of microcirculation with laser-based technique will be initiated upon the ethical consent is approved. Fifty burn patients will be included in the study. All patients will be asked for the existence of any comorbid disease. Once the patient meets the inclusion criteria, he will be eligible for the study.

LSCI and LDI devices will alternately be used to record blood flux. Burn wound including the healthy area 5 cm wider than the borders will be scanned by LDI and LSCI. After completing the data collection, all images will be compared to test the linearity between arbitrary units of LDI and LSCI. Based on the measured blood flux, a color image will be created, based on a color map created in a study on volunteers. Blood flux is calculated by the dedicated software.

Names of the patients will be coded with numbers. Only the main investigator will be aware of who corresponds to which number. Results of Perimed (LSCI) and Moore Devices (LDI) will be analyzed with the software PIMsoft 1.5 (Perimed AB, Järfälla, Sweden), MoorLDI2-BI Burn's Software Version 4.0, respectively. Two investigators will perform the analysis. If one investigator will make the analysis, the other will check the results, as well. Stored data will be extracted and stored coded in the castor study management system en electronic data capture system.

Assessment of microcirculation with the Perimed LSCI Pericam PSI System (Perimed AB, Järfälla, Sweden) Laser Speckle Contrast Imager is used to measure skin perfusion. The system uses a divergent laser beam with a wavelength of 785 nm. Perfusion images are acquired by averaging data from 21 images taken in rapid succession (acquisition time 1 seconds), over 1-minute intervals. A flexible working distance from 10 to 40 cm allows measurement areas up to 24 x 24 cm. Tissue blood perfusion is visualized in real time with a resolution of up to 100 µm/pixel. The system is calibrated according to the manufacturer recommendations. Perfusion images will be further analyzed by calculating mean perfusion levels in regions of interest using PIMsoft 1.5 (Perimed AB, Järfälla, Sweden).

Operating procedures:

1. Switch on the computer and any peripherals
2. Switch on the Perimed instrument to be used via the switch on the rear panel
3. Allow the instrument at least 5 minutes for warm-up
4. Start the PIMSoft software on computer
5. Make sure that you allowed the subject at least 20 minutes to rest and acclimatize before the measurement, make sure the subject is in a comfortable position.
6. Position the instrument head within the recommended measurement distance from the tissue (10-40 cm)
7. The head should be parallel, and the laser beam perpendicular to the tissue being measured
8. Set the size of the measurement area by entering the desired width and height in the corresponding text boxes. Select a point density (resolution).
9. Click on the start button
10. After recording the image and/or video click on the stop button and finalize the recording
11. Recorded document is already saved to the computer

Assessment of microcirculation with the Moor LDI

MoorLDI2-BI System (Moor Instruments Ltd., Axminster, Devon, UK) is used to measure skin perfusion. The system uses a divergent laser beam with a wavelength of 633 nm. A flexible working distance from 30 to 100 cm allows measurement areas up to 50 x 50 cm. Scan times are ranging from 40 seconds up to 2 minutes. The scan speed is approximately 4ms/pixel. Tissue blood perfusion is visualized in real time with a maximum image resolution of 256x256 pixels. The system is calibrated according to the manufacturer recommendations. Perfusion images will be further analyzed by calculating mean perfusion levels in regions of interest using MoorLDI2-BI Burn's Software Version 4.0.

Operating procedures:

1. It is common practice to perform moorLDI2-BI scans after dressings have been removed during routine dressing change. This avoids extra patient discomfort.
2. Remove dressings (during routine wound management) and any cream (e.g., silver sulphadiazine) to a light smear or better.
3. Position the patient with due regard to maintenance of a sterile environment for the wound. The wound should be held in a comfortable position so that it can be held reasonably still for the duration of the moorLDI2-BI scan.
4. The patient should breathe normally during the scan and should avoid coughing or holding breath.
5. When scanning the face and/or upper body areas, the eyes must be covered. If the patient is unable to wear eye protection, the face must not be scanned.
6. Ensure that the room or space to be used for scanning has the correct laser warning labels and screening
7. Ensure clean or sterilized eye protection is on hand for patient and staff if required.
8. Angle the scan head downwards prior to turning on the moorLDI2-BI.
9. Turn on the moorLDI2-BI.
10. Enter Patient Information; use the Comment box for details of sickness, medication or any other factors which may influence peripheral blood flow.
11. Plan to avoid scanning under direct sunlight, theatre lights or another bright lighting.
12. Plan the scan head positions for all burn wounds. Consider scan directions that will avoid direct reflection of the moorLDI2-BI laser back into the scan head from moist wound surfaces.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 16 years old
* Acute burn wounds admitted in the Burn Centre of the Maasstad hospital
* Assessment burn wounds with laser Doppler imager

Exclusion Criteria:

* Pregnant
* Unconscious patients

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: • All consecutive adult patients with acute burn wounds, who are seen within 5 day post burn in the Burn Centre of the Maasstad hospital are eligible to enroll in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
primary outcome | 10 minutes
  o To validate the LSCI device (Perimed AB, Järfälla, Sweden) in burn patients.

SECONDARY OUTCOMES:
secondary outcome | 10 minutes
  o To validate a color code, comparing LDI (moorLDI2-Burn Imager™ (Moor Instruments, Axminster, United Kingdom) and LSCI in burn patients

CONTACTS AND LOCATIONS:
Locations (1):
- Maastad hospital, Rotterdam, South Netherlands, Netherlands

IPD SHARING:
Plan to Share IPD: No